CLINICAL TRIAL: NCT00199342
Title: An Open-Label Study of KW-2871 Administered With a Premedication Regimen in Patients With Advanced Stage IV Melanoma
Brief Title: A Study of a Monoclonal Antibody, KW-2871, in Patients With Advanced Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Occurrence of 2 dose-limiting toxicities at the initial dose level (60 mg/m2) in Part I.
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Kent Allenby, MD/Consultant, Kyowa Hakko Kirin Pharma, Inc
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2871-US-002
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Stage IV Melanoma
Keywords: Melanoma; Monoclonal Antibody; Anti-GD-3
MeSH Terms: conditions — Melanoma | interventions — ecromeximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: KW-2871 — potentially therapeutic monoclonal antibody for the treatment of advanced stage four melanoma

SUMMARY:
This is a dose escalating cohort study to determine the maximum tolerated dose (MTD) of KW-2871 (in dose cohorts of 60, 80, and 100 mg/m2) when administered with a specified premedication regimen (ranitidine, diphenhydramine, and dexamethasone). KW-2871 will be administered at 14-day intervals.

DETAILED DESCRIPTION:
This open label study consists of two parts. Part I, the Phase I component of the study, will be conducted at a single center, and will enroll up to 18 patients with histologically documented Stage IV melanoma (per the American Joint Committee on Cancer [AJCC] criteria) that is not currently amenable to surgical resection or other therapies.

A specified premedication regimen consisting of ranitidine, diphenhydramine, and dexamethasone will be administered to all patients 30 minutes prior to infusion of any dose of KW-2871.

Planned doses of KW-2871 are 60 mg/m2, 80 mg/m2, 100 mg/m2

After identification of the MTD, 30 patients will be enrolled at that dose level in Part II of the study. If no MTD is identified after treatment with the 100 mg/m2 dose level, the dose administered in Part II of the study will be 100 mg/m2. If the MTD is determined as 60 mg/m2, this study will be closed to further patient accrual and will not proceed to Part II.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years of age
2. Patients with documented Stage IV melanoma (histologically- or cytologically-proven, as per AJCC criteria) that is not currently amenable to surgical resection (due to either medical contraindication or non-resectability of tumor)
3. Patients may have measurable or non-measurable disease, in accordance with the RECIST criteria.
4. Failure of at least one, but no more than 3, standard treatment regimen(s) for metastatic disease
5. Patients must have adequate end-organ function including:

   1. Hemoglobin > 9.0 g/dL
   2. ANC > 1500/mm3
   3. Platelet count > 100,000/ mm3
   4. Serum creatinine < 1.5x the upper limit of normal
   5. Total bilirubin < 1.5 mg/dL
   6. AST or ALT < 3 X the upper limit of normal
   7. Serum albumin > 2.5 g/dL
6. Patients with an ECOG performance status of 0, 1, or 2, and an expected survival of > 12 weeks
7. Patients must be able to provide written informed consent (must be obtained at time of patient screening)
8. Female patients of childbearing potential must not be pregnant or breast-feeding and must have a negative serum pregnancy test within 72 hours prior to administration of the first dose of KW-287. Women are NOT considered of child-bearing potential after surgical sterilization with physician-documented hysterectomy or tubal ligation, or if post-menopausal; post-menopausal status is defined as absence of menses for at least two consecutive years and a serum FSH > 30 IU/L in the absence of hormone replacement therapy
9. At least four weeks from last dose of systemic chemotherapy (6 weeks if mitomycin C or a nitrosourea) and recovery from any acute toxicity
10. At least four weeks from last radiotherapy treatment, with recovery from any acute toxicity

Exclusion Criteria:

1. Women who are pregnant or lactating and women of childbearing potential and fertile men not agreeing to a medically effective method of contraception. Women of childbearing potential will be informed as to the potential risk of procreation while participating in this study and will be advised that they must use effective contraception (e.g. oral contraceptive or long-term injectable or implantable hormonal contraceptive, double-barrier methods such as condom and diaphragm, condom and foam, condom and sponge or intra-uterine devices) during the treatment period and for a period of 3 months following the completion of dosing.
2. Patients with significant cardiovascular disease as defined by The New York Heart Association Classification (Class III or higher)
3. Patients with symptomatic or known brain metastases unless patient has undergone radiotherapy (or treatment with gamma knife) or resection of an isolated lesion and maintenance steroids are not required
4. Patients with a history of another malignancy within the last 2 years with the exception of:

   * Treated, non-melanoma skin cancers
   * Carcinoma in situ of the breast or cervix
   * History of T1a or b carcinoma of the prostate detected incidentally and comprising <5% of resected tissue, with PSA within normal limits since resection
5. Patients with any uncontrolled infection or other intercurrent illness
6. Patients with any history of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of an underlying disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications
7. Patients with known HIV infection
8. Patients with inadequate recovery from any prior surgical procedure
9. Patients with psychiatric disorders or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies
10. Patients with any prior monoclonal antibody therapy for melanoma
11. Patients previously treated with any other immunotherapy, vaccine, or biological response modifier therapy for melanoma, either during or within four weeks prior to study entry
12. Patients with systemic hormonal therapy, either during or within four weeks prior to first dose of KW-2871, unless for appetite stimulation
13. Patients requiring maintenance systemic steroid therapy for any condition

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-11; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To determine the MTD and a recommended Phase II dose of KW-2871 administered with a specified premedication regimen (rantidine, diphenhydramine, and dexamethasone) in patients with Stage IV melanoma. | up to 1 year
  Until determination of MTD or recommended dose for evaluation

SECONDARY OUTCOMES:
To characterize the safety and tolerability profile of KW-2871 when administered with a specified premedication regimen. | up to 1 year
To obtain a preliminary assessment of antineoplastic activity of KW-2871, as measured by the number of objective antitumor responses, duration of response, time to progression (TTP) and survival in this patient population. | up to 1 year
To characterize the pharmacokinetic profile of indicated dose levels of KW-2871 when administered with this specified premedication regimen. | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero, MD, Principal Investigator — Comprehensive Cancer Center University of Alabama
Locations (2):
- United States (2):
  - Comprehensive Cancer Center- University of Alabama at Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center, Tampa, Florida